CLINICAL TRIAL: NCT02139527
Title: The Centers for Arthroplasty Research and Education in Spine (CARES) Lumbar Artificial Disc Registry Protocol
Brief Title: CARES Lumbar Artificial Disc Registry
Status: Terminated | Type: Observational
Why Stopped: Low enrollment and follow-up data on enrolled patients.
Sponsor: DePuy Spine (Industry)
Responsible Party: Sponsor
Other Study IDs: 06-CAD-01
Record Dates: First submitted 2014-02-11; First posted 2014-05-15 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Lumbar Degenerative Disc Disease
Keywords: arthroplasty; spinal; CHARITE; PRODISC-L; PRODISC; disc; replacement; lumbar
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Total Disc Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Total Disc Replacement
  Other Names: CHARITE™ Artificial Disc; PRODISC®-L Total Disc Replacement

SUMMARY:
The purpose of the registry is to assess outcomes following treatment with lumbar total disc replacement (TDR) in patients outside the clinical trial setting.

DETAILED DESCRIPTION:
The purpose of this study is to capture outcomes associated with use of total disc replacement (TDR) in patients treated with either the CHARITE™ Artificial Disc or the PRODISC®-L Total Disc Replacement may be included in the registry.

ELIGIBILITY:
Key Inclusion Criteria:

* Treated with the lumbar TDR.
* Signed IRB approved consent document.

Key Exclusion Criteria:

* None known.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that undergo lumbar total disc replacement (TDR); this includes patients treated with either the CHARITE disc or the ProDisc-L disc
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index (ODI) Score | 3, 6, 12, 24, 36, 48, and 60 months post operative
  The ODI assesses several domains of function affected by low back pain. A change of 15 points from baseline is considered a clinical meaningful difference for the individual. The change from pre operative baseline to each follow-up assessment will be calculated.